CLINICAL TRIAL: NCT02316431
Title: Diagnostic Comparison and Workflow Evaluation of Whole Body PET-magnetic Resonance and PET-CT With and Without Contrast Media in Patients With Oncologic Diseases
Brief Title: Diagnostic Comparison of PET-magnetic Resonance and PET-CT in Patients With Oncologic Diseases
Acronym: Workflow
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr. 2014-0072
Record Dates: First submitted 2014-12-09; First posted 2014-12-12 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Neoplasm Staging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Diagnostic accuracy of PET/magnetic resonance and PET/CT will be compared concerning primary tumor, regional nodes, metastasis (TNM) staging and therapeutic influence. Workflow scenarios will be evaluated to create imaging protocols which are time efficient and diagnostically accurate.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients from 18-90 years
* Written informed consent
* Patients with a proven or suspected oncological disease referred for a clinically -Indicated PET/CT with of without contrast media

Exclusion Criteria:

* Pregnant or breast feeding women
* Non compliance of the patient to follow the study instructions (e.g. hearing problems, dementia)
* Inclusion in another clinical trial 30 days prior to inclusion
* Age < 30years
* Contraindication for MRI (cardiac pacemaker, certain metal implants, claustrophobia
* Known allergies to contrast CT or MRI contrast media
* Patients with an glomerular filtration rate of < 60ml/min/1.73m2

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a proven or suspected oncological disease referred for a clinically indicated PET/CT with of without contrast media.
Sampling Method: Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2014-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with correct TNM staging defined with PET/magnetic resonance versus PET/CT | 12 month

SECONDARY OUTCOMES:
Number of minutes needed per PET/magnetic resonance protocol compared to PET/CT | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Veit-Haibach, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Diagnostic and Interventional Radiology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Sekine T, Delso G, Zeimpekis KG, de Galiza Barbosa F, Ter Voert EEGW, Huellner M, Veit-Haibach P. Reduction of 18F-FDG Dose in Clinical PET/MR Imaging by Using Silicon Photomultiplier Detectors. Radiology. 2018 Jan;286(1):249-259. doi: 10.1148/radiol.2017162305. Epub 2017 Sep 14. PMID 28914600